CLINICAL TRIAL: NCT01456481
Title: Assessment of Midodrine in the Prevention of Vasovagal Syncope: The Prevention of Syncope Trial IV (Post 4)
Brief Title: Assessment of Midodrine in the Prevention of Vasovagal Syncope: The Prevention of Syncope Trial IV
Acronym: POST 4
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Bob Sheldon (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor-Investigator, Dr. Bob Sheldon, Professor of Cardiac Sciences, Medicine and Medical Genetics, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIHR#243314
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Vasovagal Syncope
Keywords: reflex fainting; vasovagal syncope; midodrine
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midodrine hydrochloride pills (Active Comparator)
  Interventions: Drug: midodrine hydrochloride
- oral placebo or sugar pill (Placebo Comparator)
  Interventions: Drug: midodrine hydrochloride; Drug: matching placebo

INTERVENTIONS:
Drug: midodrine hydrochloride — Target dose is midodrine hydrochloride or placebo pills 10 mg three times a day for 12 months. The starting dose is 5mg q4h x3, and if tolerated a forced titration up to 10mg/dose. If there is an intolerance, then the dose can be reduced to 2.5mg/dose.
  Other Names: Brand name for the drug is midodrine.
Drug: matching placebo — The target dose in this study is 10mg q4h x3 for 12 months. The starting dose is 5mg q4h x3, and if tolerated a forced titration up to 10mg/dose. If there is an intolerance, then the dose can be reduced to 2.5mg/dose.
  Arms: oral placebo or sugar pill

SUMMARY:
About 20% of adults faint recurrently. These patients are often highly symptomatic, have problems with employment and driving and have reduced quality of life. There are no therapies that have withstood the test of adequately designed and conducted randomized clinical trials. Midodrine is a prodrug whose metabolite is an alpha-1 adrenergic agonist that increases venous return to the heart and raises blood pressure. There is considerable lower level evidence that it might prevent vasovagal syncope.

The investigators will test the hypothesis that Midodrine prevents recurrences of syncope in patients with moderate to severe vasovagal syncope.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have:

  * ≥2 syncopal spells in the year preceding enrolment, and
  * ≥ -2 points on the Syncope Symptom Score for Structurally Normal hearts, and
  * Age ≥ 18 years with informed consent.

Exclusion Criteria:

* Patients will be excluded if they have:

  * other causes of syncope, such as ventricular tachycardia, complete heart block, postural hypotension or hypersensitive carotid sinus syndrome,
  * an inability to give informed consent,
  * important valvular, coronary, myocardial or conduction abnormality or significant arrhythmia,
  * hypertrophic cardiomyopathy,
  * a permanent pacemaker,
  * a seizure disorder,
  * urinary retention,
  * hypertension defined as >140/90 mm Hg,
  * hepatic disease,
  * glaucoma or
  * a 5-minute stand test resulting in diagnoses of Postural Orthostatic Tachycardia Syndrome or Orthostatic Hypotension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-11; Primary Completion 2018-12-20 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the proportion of patients having at least one syncope recurrence. | 1 year.

SECONDARY OUTCOMES:
A secondary outcome will be the time between the first and second syncope recurrences. | 1 year
A secondary outcome will be the frequency of syncopal spells. | 1 year
A secondary outcome is the number, duration, and severity of presyncopal spells (as measured with the Calgary Presyncope Scale(19)). | 1 year.
A secondary outcomes will be quality of life as measured by the EQ-5D and the ISQL. | 1 year

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Vanderbilt University, Nashville, Tennessee
- Canada (14):
  - University of Calgary, Calgary, Alberta
  - Alberta Health Services - Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Victoria Cardiac Arrythmia Trials, Victoria, British Columbia
  - St. Boniface General Hospital, St. Boniface, Manitoba
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - Queen E II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Hopital Sacre Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Prairie Vascular Research Network/Regina General Hospital, Regina, Saskatchewan
  - Saskatoon Cardiology Consultants/Royal University Hospital, Saskatoon, Saskatchewan
- Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Derived] Sheldon R, Faris P, Tang A, Ayala-Paredes F, Guzman J, Marquez M, Morillo CA, Krahn AD, Kus T, Ritchie D, Safdar S, Maxey C, Raj SR; POST 4 investigators. Midodrine for the Prevention of Vasovagal Syncope : A Randomized Clinical Trial. Ann Intern Med. 2021 Oct;174(10):1349-1356. doi: 10.7326/M20-5415. Epub 2021 Aug 3. PMID 34339231
- [Derived] Raj SR, Faris PD, McRae M, Sheldon RS. Rationale for the prevention of syncope trial IV: assessment of midodrine. Clin Auton Res. 2012 Dec;22(6):275-80. doi: 10.1007/s10286-012-0167-5. Epub 2012 May 19. PMID 22610268